CLINICAL TRIAL: NCT06680674
Title: Multinational Cross-sectional Review of Diabetes and Obesity Management in Hospitals Across Europe: The DIABESITY Survey
Brief Title: Multinational Point Prevalence Study on the Management of Diabesity in Hospitals
Acronym: DiabesityDay
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Hospital de Cascais Dr. José de Almeida (Portugal) (Unknown); Centre Hospitalier Universitaire Sétif, Service Médecine Interne (Algeria) (Unknown); Rabin Medical Center (Other); Hospital Regional de Malaga (Other); Charles University, Czech Republic (Other); University Hospital Bratislava (Other); Complejo Hospitalario de Especialidades Juan RamÃ³n Jimenez (Unknown); Medical University Innsbruck (Other); Aristotle University Of Thessaloniki (Other); Rostov State Medical University (Unknown); Hospital Marina Baixa (Unknown); Riga East Clinical University Hospital (Other Government); University Hospital, Aachen (Other); San Raffaele University Hospital, Italy (Other); Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ann-Kristin Porth, Research Assistant (PhD), Medical University of Vienna
Other Study IDs: EK 1828/2024
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine care for people with diabetes, with or without obesity, in the hospital setting — Routine care for people with diabetes, with or without obesity, in the hospital setting, including routine pharmacological treatment for diabetes and obesity.

SUMMARY:
Diabetes related to obesity ("diabesity") is becoming increasingly prevalent. Hospitalizations among people with diabetes are frequent and glycaemic control is often suboptimal during these stays.

However, the pharmacological treatment of diabesity has made significant progress in recent years.

The objective of this study is to assess the management of diabesity in the international hospital setting. Aims include:

1. to determine the prevalence of causes and duration of hospitalization
2. to investigate the treatments used
3. to determine individual metabolic control achived This is a cross-sectional multi-centre study in which researchers will conduct a one-day point prevalence assessment in internal medicine wards.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the time of the survey for any cause
* Diabetes diagnosis (Known / documented in medical history or newly diagnosed using ADA diagnostic criteria)
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Patients in wards and units other than internal medicine wards (such as outpatient areas, emergency departments, skilled nursing and intensive care units, etc.)
* Paediatric patients (Age < 18 years)
* Patients without a diabetes diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age ≥ 18 years) with diabetes who are admitted to an internal medicine ward of a participating medical centre at the time of the study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of point-of-care glucose values | 3 days
  Mean number of point-of-care glucose measurements during hospitalization

SECONDARY OUTCOMES:
Severe hypoglycaemia | From day of admission to the day of data collection, i.e., November 14, 2024
  Severe hypoglycaemia during admission (glucose <40mg/dL)

OTHER OUTCOMES:
Diabetes treatment during hospitalization | From day of admission to the day of data collection, i.e., November 14, 2024
  Diabetes treatment used during the time of hospitalization
Insulin regimen during hospitalization | From day of admission to the day of data collection, i.e., November 14, 2024
  Insulin regimen used during the time of hospitalization (e.g., correction, basal, prandial bolus)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Prof, Study Director — Medical University of Vienna
Locations (8):
- Medical University of Vienna, Vienna, Austria
- General University Hospital in Prague, Prague, Czechia
- University Hospital RWTH Aachen, Aachen, Germany
- Hippokration General Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece
- Rabin Medical Center, Hasharon Hospital, Petah Tikva, Israel
- Riga East Clinical University Hospital, Riga, Latvia
- Rostov State Medical University, Rostov-on-Don, Russia
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data will only be shared in aggregated form.